CLINICAL TRIAL: NCT04383743
Title: Pembrolizumab and aMVAC Chemotherapy as Neoadjuvant Therapy in Non-Urothelial Histology Muscle-Invasive Bladder Cancer: A Pilot Trial
Brief Title: Pembrolizumab and Combination Chemotherapy Before Surgery for the Treatment of Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Petros Grivas, MD, PhD, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1006206; NCI-2019-08028 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10439 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Muscle Invasive Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Methotrexate; merphos; pegfilgrastim; pembrolizumab; Cystectomy; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, aMVAC) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of weeks 0, 3, and 6 and methotrexate IV, vinblastine IV, doxorubicin IV, and cisplatin IV on day 1 of weeks 0, 2, 4, and 6 in the absence of disease progression or unacceptable toxicity. Patients also receive pegfilgrastim SC on day 1 or 2 of weeks 0, 2, 4, and 6 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care radical cystectomy.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin; Drug: Methotrexate; Biological: Pegfilgrastim; Biological: Pembrolizumab; Procedure: Radical Cystectomy; Drug: Vinblastine Sulfate

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim-jmdb; SD-01; SD-01 sustained duration G-CSF; Nyvepria; Pegcyte; Udenyca; Ziextenzo
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Radical Cystectomy — Undergo standard of care radical cystectomy
  Other Names: Complete Cystectomy
Drug: Vinblastine Sulfate — Given IV
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE

SUMMARY:
This pilot study is evaluating how well pembrolizumab and combination chemotherapy before surgery work for the treatment of specific types of muscle-invasive bladder cancer that have unusual appearance (variants). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as methotrexate, vinblastine, adriamycin, and cisplatin work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab and combination chemotherapy before surgery may work better in treating patients with these muscle invasive bladder cancer variants compared to chemotherapy alone.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of weeks 0, 3, and 6 and methotrexate IV, vinblastine IV, doxorubicin IV, and cisplatin IV on day 1 of weeks 0, 2, 4, and 6 in the absence of disease progression or unacceptable toxicity. Patients also receive pegfilgrastim subcutaneously (SC) on day 1 or 2 of weeks 0, 2, 4, and 6 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care radical cystectomy.

After completion of study treatment, patients are followed up about 1 month after surgery and then every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diagnosis of muscle invasive bladder cancer (cT2-T4a, N0-N1, M0 clinical stage per American Joint Commission on Cancer [AJCC]). Clinical node-positive (N1) patients are eligible provided the lymph nodes (LNs) are confined to the true pelvis and are within the planned surgical LN dissection template
* Histology must be either pure or predominant non-urothelial histology (noted on any TURBT)
* Participants must be deemed eligible for cisplatin-based chemotherapy, radical cystectomy (RC) and pelvic lymph node dissection (PLND) by urologist and medical oncologist
* Patients must agree to undergo curative intent surgery
* TURBT that showed muscularis propria invasion should be within 12 weeks prior to beginning study therapy. Patients must have available tumor tissue from either initial or repeat TURBT, prior to starting study therapy. Archival tumor tissue sample of a tumor lesion (TURBT specimen) should be provided and must contain muscle invasive component, at least >= T2 tumor. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory, preferably within 14 days from the date slides are cut if possible. Patient must be willing to provide tumor tissue for research. Research samples will not be used for any studies unrelated to this trial
* Must have clinical non-metastatic bladder cancer (M0) determined by cross-sectional computed tomography (CT) chest, abdomen and pelvis (CAP) or magnetic resonance imaging (MRI) imaging
* A male participant must agree to use a contraception during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant , not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 180 days after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. Evaluation is to be performed within 7 days prior to the date of enrollment
* Absolute neutrophil count (ANC) >= 1500/uL (collected within 10 days prior to the start of study treatment)
* Platelets >= 100 000/uL (collected within 10 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (collected within 10 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Serum creatinine =< 1.5 x upper limits of normal (ULN) OR calculated creatinine clearance (glomerular filtration rate [GFR] can be used in place of creatinine or creatinine clearance) >= 50 ml/min (collected within 10 days prior to the start of study treatment). Measured or calculated creatinine clearance (GFR can be used in place of creatinine clearance; 24-hour urine collection can be used for more accurate estimate as needed)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (collected within 10 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (collected within 10 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy, as long as PT is within therapeutic range of intended use of anticoagulants (collected within 10 days prior to the start of study treatment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy, as long as aPTT is within therapeutic range of intended use of anticoagulants (collected within 10 days prior to the start of study treatment)

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Patients with pure small cell histology will be excluded. Mixed histology including partial neuroendocrine small cell features will be permitted
* Patients considered to be medically unfit for accelerated (dose dense) MVAC chemotherapy, TURBT or RC (per investigator discretion) will be excluded
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks. Intravesical therapies are allowed without specified treatment interval

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. If participant had major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and should not have active radiation pneumonitis
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, a version of varicella/zoster (chicken pox), yellow fever, rabies, Bacillus calmette-guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing > 10 mg daily of prednisone dose equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has known additional malignancy that is progressing or has required active systemic treatment within the past 2 years. Note: Participants with basal cell carcinoma or squamous cell carcinoma of the skin, or any carcinoma in situ that have undergone potentially curative therapy are not excluded. Low/intermediate risk prostate cancer with prior potentially curative therapy, or no intent of future systemic therapy and/or radiation is allowed. Non-invasive (Tis, Ta) upper urinary tract (renal pelvis/ureter) is allowed. Urethra cancer with prior curative intent therapy with no active recurrence is also allowed regardless of time elapsed
* Has known locally advanced (unresectable) or metastatic cancer on baseline radiographic imaging (CT or MRI) obtained within 28 days prior to study registration
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed. Note: Patients with active well controlled type 1 diabetes mellitus, vitiligo, Graves' disease, Hashimoto disease, eczema, lichen simplex chronicus, or psoriasis, not requiring systemic immunosuppression within the past 2 years are not excluded
* Has history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has known history of human immunodeficiency virus (HIV). Note: no HIV testing is required
* Has known history of active hepatitis B (defined as hepatitis B surface antigen [HBsAg] detected) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] detected) infection. Note: no testing for hepatitis B and hepatitis C is required
* Has known history of active TB (Bacillus tuberculosis). Note: no testing is required unless it is clinically indicated
* Has history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has had allogeneic solid visceral organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petros Grivas, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Percentage of patients with no histologic evidence of tumor at time of cystectomy (ypT0N0)
Time Frame: At time of radical cystectomy at approximately within 10 weeks of last neoadjuvant infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Number analyzed (Participants) | 17
Participants | 9

2. Secondary Outcome: Frequency of Any Adverse Event According to Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) Related to Study Therapy.
Description: The frequency of toxicity of study therapy regimen. Measured as the number of participants that experienced an AE (any grade) related to study therapy while on trial.
Time Frame: Up to 90 days post study therapy completion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Number analyzed (Participants) | 17
Participants | 17

3. Secondary Outcome: Frequency of Grade 3 or Greater Adverse Events According to Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) Related to Study Therapy.
Description: The severity of toxicity of therapy regimen. Measured as the number of participants that experienced an AE of grade 3 or higher related to study therapy while on trial
Time Frame: Up to 90 days post therapy completion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Number analyzed (Participants) | 17
Participants | 8

4. Secondary Outcome: Estimated 2-year Event-free Survival (EFS)
Description: Percentage reported represents an estimate using the method of Kaplan-Meier 2-year EFS Estimate (95% CI)
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Number analyzed (Participants) | 17
percentage of participants | 64 [32 to 84]

5. Secondary Outcome: Number of Participants Able to Undergo Radical Cystectomy Within 10 Weeks From Completion of Study Therapy
Description: To evaluate the feasibility of neoadjuvant aMVAC and pembrolizumab as measured by the rate of patients able to receive RC within 10 weeks from completion of study therapy
Time Frame: within 10 weeks from completion of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, aMVAC)
Number analyzed (Participants) | 17
Participants | 14

6. Other Pre Specified Outcome: Tumor Infiltrating Lymphocyte (TIL) Density
Description: TIL density will be summarized by means, medians, and quantiles. Changes will be evaluated as both absolute and percentage change. Descriptive statistics will also be used when needed.
Time Frame: At time of Transurethral Bladder Tumor Resection and radical cystectomy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Pembrolizumab, aMVAC)
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, aMVAC) (N=17)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (4)
Kidney Infection (Infections and infestations) | 3 (4)
Fever (General disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, aMVAC) (N=17)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 9 (30)
Anorexia (Metabolism and nutrition disorders) | 9 (14)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Concentration Impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine Increased (Investigations) | 4 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (5)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 8 (9)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 11 (11)
Fever (General disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot Flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (7)
Hypotension (Vascular disorders) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 7 (9)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (17)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Periodontal Disease (Gastrointestinal disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet Count Decreased (Investigations) | 3 (4)
Presyncope (Nervous system disorders) | 1 (2)
Respiratory, Thoracic and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial Thrombophlebitis (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 6 (6)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Vision Decreased (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 2 (6)
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 (4)
Allergic Reaction (Immune system disorders) | 1 (2)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 3 (3)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Bladder Infection (Infections and infestations) | 1 (4)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Metabolism and Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1 (1)
Neoplasms Benign, Malignant and Unspecified (Incl Cysts and Polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04383743/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04383743/ICF_000.pdf